CLINICAL TRIAL: NCT02012270
Title: Prospective Case-control Study on the Incidence of Incisional Hernias at 12 Months After Closure of Midline Laparotomies in Patients Treated for Abdominal Aortic Aneurysm
Brief Title: Aneurysma Hernia Study - Incidence of Incisional Hernias After Abdominal Aortic Aneurysm Repair
Acronym: АНЕУРИЗМА
Status: Completed | Type: Observational
Sponsor: Igor Koncar (Other)
Collaborators: University Hospital, Ghent (Other); Medical University of Gdansk (Other)
Responsible Party: Sponsor-Investigator, Igor Koncar, Igor Koncar, University of Belgrade
Organization: University of Belgrade (Other)
Other Study IDs: 175008
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Incisional Hernia; Abdominal Aortic Aneurysm
Keywords: Aortic Aneurysm; Hernia; Abdominal Wound Closure Techniques
MeSH Terms: conditions — Incisional Hernia; Aortic Aneurysm, Abdominal; Aortic Aneurysm; Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional Group: Group of patients in whom after open AAA repair abdominal wall will be closed by conventional technique by the operating surgeons. There will be a great variation in sutures and techniques used
  Interventions: Procedure: Conventional group
- PRINCIPLES Group: Group of patients in whom after open AAA repair abdominal wall will be closed by PRINCIPLES technique by the operating surgeons.
  Interventions: Procedure: PRINCIPLES technique

INTERVENTIONS:
Procedure: PRINCIPLES technique — Principles technique for closure of midline laparotomy incisions
  * closure with a running suture of a slowly absorbable monofilament suture- Monomax 2/0 of 150 cm length with a taper needle point ((1/2 circle, size: 30mm) (B.Braun, reference 0041453)
  * the suture is started and ended with a self-locking knot, if more than one suture is used sutures are knotted separately, only the fascia will be sutured with small stitches close to each other
  * the SL/WL ratio should be at least 4/1
  * SL/WL = (150cm x number of sutures used) - (the suture remnants)
  * the mean stitch length should be less than 4 cm (suture length / number of stitches placed)
  Groups: PRINCIPLES Group
Procedure: Conventional group — the fascia will be closed with the current method by the surgeons. There will be a great variation in sutures and techniques used. Study group: the fascia will be closed according
  Groups: Conventional Group

SUMMARY:
Principles= Prevention of incision hernias by primary closure of mid line laparotomies with the best-evidenced suture techniques.

Background:

Surgical practice of abdominal wall closure continues to rely largely on tradition rather than high-quality level I evidence. Incisional hernia after laparotomy for treatment of abdominal aortic aneurysm (AAA) has a high incidence.

At this moment the best results in a prospective randomised clinical trial considering incision hernia rates and wound infections, have been reported by the surgeons from the Sundsvall clinic in Sweden. Their technique using a suture to wound length ratio of at least 4/1 and using many small stitches will be described in the protocol as the "Principles Technique". We want to explore if these results can indeed prevent incision hernias significantly if implemented with training and tutoring.

Methodology:Vascular surgeons,who are not using the principles yet, but show an interest to learn the Principles, will be asked to monitor a cohort of AAA patients using their current sutures and surgical techniques. Some of the vascular surgeons will undergo training and if wanted, proctoring during the first procedures using the Principles. A cohort of 120 AAA patients will be closed according to the Principles and monitored. The results of these 120 patients will be compared to the control group consisting of patients closed with the conventional technique by non---trained surgeons. Primary endpoint:The incidence of incision hernias at 12 months will be determined by clinical examination.

Data management and ownership:

The data will be collected on a paper form and will be introduced is a database (SPSS Statistics, IBM) from which statistical analysis will be made.

DETAILED DESCRIPTION:
Principles= Prevention of incision hernias by primary closure of mid line laparotomies with the best-evidenced suture techniques.

Background:

Although many data from prospective studies have set some evidence-based principles to be adopted when closing mid line laparotomy incisions, these principles have not found a widespread implementation in the surgical community. Surgical practice continues to rely largely on tradition rather than high-quality level I evidence. Incision hernia after laparotomy for treatment of abdominal aortic aneurysm (AAA) has a high incidence of 10% to 37% depending on the method of follow up (clinically, with ultrasound or with CT scan) and the duration of follow up.

It is known that the surgical technique used to close the fascia in mid line laparotomies is an important parameter with regard to wound complications like wound infections and incision hernias. At this moment the best results in a prospective randomised clinical trial considering incisional hernia rates and wound infections, have been reported by the surgeons from the Sundsvall clinic in Sweden. Their technique using a suture to wound length ratio of at least 4/1 and using many small stitches will be described in the protocol as the "Principles Technique". We want to explore if these results can indeed prevent incision hernias significantly if implemented with training and tutoring.

Methodology:Vascular surgeons,who are not using the principles yet, but show an interest to learn the Principles, will be asked to monitor a cohort of AAA patients using their current sutures and surgical techniques. Some of the vascular surgeons will undergo training and if wanted, proctoring during the first procedures using the Principles. A cohort of 120 AAA patients will be closed according to the Principles and monitored. The results of these 120 patients will be compared to the control group consisting of patients closed with the conventional technique by non---trained surgeons. Study hypothesis and sample size calculation: Investigators might improve the incision hernia rate after AAA treatment through a mid line incision at 12 months by using the Principles from an estimated 25% in the conventionally closed patients to 10% in the patients closed using the Principles.

Calculation:

To show a decrease of 60% in the incision hernia rate at 12 months(25% vs 10% incision hernias at 12 months)with a power of 80% and a significance level of 5%, investigators need 100 evaluable patients at 12 months in each arm. To compensate a 20% lost to follow up, we have to include at least 120 patients before the "principles training" and 120 patients afterwards. So the trial will end inclusions when 120 AAA patients have been entered using the Principles. Most likely the control group will be larger than these 120 patients,depending on the number of vascular surgeons participating in the teaching course and the timing of this course.

Primary endpoint:The incidence of incision hernias at 12 months will be determined by clinical examination.

Data management and ownership:

The data will be collected on a paper form and will be introduced in a database (SPSS Statistics, IBM) from which statistical analysis will be made.

ELIGIBILITY:
Inclusion Criteria:All patients undergoing treatment for an abdominal aortic aneurysm in the department of vascular surgery at the Serbian Clinical Centre in Beograd, Serbia, through midline laparotomies are eligible for the trial.

Exclusion Criteria:

patients not willing to take part in the follow up visits after informed consent no other exclusion criteria will be used (emergency, previous laparotomy or hernia repair)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient operated due to Abdominal Aortic Aneurysm with open repair through laparotomy.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The incidence of incisional hernias | 12 months
  Incidence of incisional hernia after AAA repair after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lazar Davidovic, Prof, Principal Investigator — University of Belgrade; Zivan Maksimovic, Prof, Principal Investigator — University of Belgrade; Filip Muysoms, MD, Principal Investigator — University Ghent
Locations (2):
- Medical University of Gdansk Dept. of Cardiac and Vascular Surgery, Gdansk, Poland
- Clinic for Vascular and Endovascular Surgery, Serbian Clinical Centre, Belgrade, Serbia